CLINICAL TRIAL: NCT00025116
Title: A Randomized Phase II Study Of ZD1839 (IRESSA) In Patients With Hormone Refractory Prostate Cancer
Brief Title: ZD 1839 in Treating Patients With Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I140; CAN-NCIC-IND140 (Other: PDQ); CDR0000068915 (Other: PDQ)
Record Dates: First submitted 2001-10-11; First posted 2003-09-17 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Biological therapies such as ZD 1839 may interfere with the growth of tumor cells and slow the growth of prostate cancer. It is not yet known which dose of ZD 1839 is more effective in treating prostate cancer that has not responded to hormone therapy.

PURPOSE: Randomized phase II trial to compare different doses of ZD 1839 in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of 2 different doses of ZD 1839, in terms of objective response, PSA response, and duration of response, in patients with hormone-refractory adenocarcinoma of the prostate.
* Compare the tolerability and quantitative toxicity of these regimens in these patients.
* Determine whether there is an association between any response or stable disease and clinical benefit as assessed by changes in quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to measurable disease (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral, low-dose ZD 1839 twice daily on day 1 and once daily on days 2-28 during course 1 and then once daily on days 1-28 during subsequent courses.
* Arm II: Patients receive oral, high-dose ZD 1839 as in arm I. Treatment in both arms continues every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at the end of each course during study, and then at 4 weeks after study.

Patients with stable or responding disease are followed at 4 weeks and then every 3 months until disease progression. All other patients are followed at 4 weeks only.

PROJECTED ACCRUAL: A total of 30-60 patients (15-30 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* PSA at least 20 ng/mL at study entry
* Must have documented evidence of disease progression, defined by 1 of the following conditions:

  * Rising PSA documented after discontinuation of peripheral antiandrogens

    * Minimum evidence of progression is a 25% increase in PSA over the reference value, provided that the increase is at least 5 ng/mL

      * Must have a first increase in PSA documented at least 1 week after the reference value and a second increase in PSA documented at least 1 week after the first increase
  * Progressive measurable disease during androgen ablative therapy (including medical or surgical castration)
* Castrate level (no greater than 50 ng/mL) of testosterone required if receiving medical androgen-ablative therapy at study entry
* Concurrent luteinizing hormone-releasing hormone agonist therapy required if receiving this medication at study entry

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN (5 times ULN if documented liver metastases)

Renal:

* Creatinine no greater than 2 times ULN

Other:

* No other malignancy within the past 5 years
* No active uncontrolled bacterial, fungal, or viral infection
* No significant neurological disorder that would preclude informed consent
* No other serious illness or medical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Concurrent epoetin alfa allowed

Chemotherapy:

* No prior chemotherapy
* No concurrent cytotoxic therapy

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior peripheral antiandrogens (6 weeks for bicalutamide)
* Concurrent steroids allowed if on stable dose for at least 4 weeks before study and no dose increase planned

Radiotherapy:

* At least 4 weeks since prior radiotherapy except low-dose, nonmyelosuppressive radiotherapy approved by the National Cancer Institute of Canada, Clinical Trials Group

Surgery:

* See Disease Characteristics
* No concurrent ophthalmic surgery

Other:

* No prior investigational agents
* No other concurrent investigational therapy
* No concurrent ketoconazole
* No concurrent high-dose narcotic therapy for pain (e.g., morphine equivalent dose more than 60 mg/day)
* Concurrent bisphosphonates allowed

Ages: 16 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-04-24 (Actual); Primary Completion 2003-06-05 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J. Moore, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Ontario Cancer Institute, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Canil CM, Moore MJ, Winquist E, Baetz T, Pollak M, Chi KN, Berry S, Ernst DS, Douglas L, Brundage M, Fisher B, McKenna A, Seymour L. Randomized phase II study of two doses of gefitinib in hormone-refractory prostate cancer: a trial of the National Cancer Institute of Canada-Clinical Trials Group. J Clin Oncol. 2005 Jan 20;23(3):455-60. doi: 10.1200/JCO.2005.02.129. PMID 15659491